CLINICAL TRIAL: NCT04666012
Title: A Phase 1/2a Study (Dose Escalation, Single Center, Open, Phase 1 and Multicenter, Open, Phase 2a) to Assess the Safety and Immunogenicity of AdCLD-CoV19: A COVID-19 Preventive Vaccine in Healthy Volunteers
Brief Title: Safety and Immunogenicity Study of AdCLD-CoV19: A COVID-19 Preventive Vaccine in Healthy Volunteers
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cellid Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: AdCLD-CoV19-001
Record Dates: First submitted 2020-12-10; First posted 2020-12-14 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Group 1: low dose (Experimental): Subject will receive single dose of AdCLD-CoV19(2.5x10^10VP) as intramuscular injection.
  Interventions: Biological: AdCLD-CoV19
- Group 2: middle dose (Experimental): Subject will receive single dose of AdCLD-CoV19(5.0x10^10VP) as intramuscular injection.
  Interventions: Biological: AdCLD-CoV19
- Group 3: high dose (Experimental): Subject will receive single dose of AdCLD-CoV19(1.0x10^11VP) as intramuscular injection.
  Interventions: Biological: AdCLD-CoV19
- Group 4: selected dose (Experimental): Subject will receive single dose of AdCLD-CoV19 as intramuscular injection.
  Interventions: Biological: AdCLD-CoV19
- Group 5: selected dose (Experimental): Subject will receive single dose of AdCLD-CoV19 as intramuscular injection.
  Interventions: Biological: AdCLD-CoV19

INTERVENTIONS:
Biological: AdCLD-CoV19 — Replication-defective human adenovirus type 5/35 vector based vaccine expressing S protein of SARS-CoV-2.

SUMMARY:
This is a Phase 1/2a clinical trial to assess the safety and immunogenicity of AdCLD-CoV19 in healthy adults.

DETAILED DESCRIPTION:
Part A is conducted as dose-escalation, single-center, open-label, a Phase 1 clinical trial. Part B is conducted as multi-center, open-label, a Phase 2a clinical trial. In Part A, we assess safety in all dose groups and set suitable two doses for Part B. In Part B, we assess immune responses against SARS-CoV-2 and set suitable dose for next phase of clinical trial. DSMB will evaluate safety during the whole study period.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to agree informed consent and aged 19 to 64 years.
2. The BMI index is 18.5 kg/m2 to 30.0 kg/m2.
3. Weigh 40kg to 100kg (Part A only)
4. Able and willing to medically effective contraception during the whole study period.
5. Agreement to refrain from blood donation during the whole study period.

Exclusion Criteria:

1. Anyone deemed infected by COVID-19.
2. Determined to be a close-contact of SARS-CoV-2 confirmed case or classified to symptomatic patient of COVID-19 prior to vaccination.
3. Clinically significant abnormal ranges of laboratory measurement, ECG, Chest X-ray at screening visit.
4. Positive in HIV, HBV, HCV test at screening visit.
5. Acute fever(≥ 38℃) or suspected infectious disease, symptoms of infectious disease(cough, difficulty breathing, chills, muscle aches, headache, sore throat, loss of smell, or loss of taste, etc.) within 3 days prior to vaccination.
6. Chronic respiratory disease: Asthma, chronic obstructive pulmonary disease, active tuberculosis, latent tuberculosis under treatment.
7. Clinically significant active or any history of disease: Hepatobiliary system, kidney, central or peripheral nervous system (epilepsy, seizure, etc.), endocrine system (uncontrolled diabetes, hyperlipidemia, etc.), cardiovascular system (congestive heart failure, coronary artery disease, myocardial infarction, control Hypertension, etc.), blood tumor, urinary system, mental, musculoskeletal system, immune system (rheumatoid arthritis, systemic lupus erythematosus).
8. Immunosuppressive disease including immunodeficiency disease.
9. Scheduled to undergo any surgery during the whole study period.
10. Healthcare worker who provide medical care to SARS-CoV-2 cases or occupationally in high risk for SARS-CoV-2 exposure during the whole study period.
11. Prisoners or subjects who are compulsorily detained. (involuntary incarceration)
12. History of SARS or MERS.
13. Allergic reaction or hypersensitivity to any ingredient of AdCLD-CoV19.
14. Having hemophilia at risk of causing serious bleeding when injected intramuscularly or receiving anticoagulants.
15. Any history of malignant disease within the past 5 years.
16. History of hypersensitivity to inoculate vaccine such as Guillain-Barre syndrome.
17. History of serious adverse reaction or allergic reaction to inoculate vaccine.
18. Urticaria past 5 years prior to vaccination.
19. History of hereditary angioneurotic edema or acquired angioneurotic edema.
20. History of solid organ or bone marrow transplantation.
21. Suspected or a history of drug or alcohol abuse past 12 month before vaccination.
22. Receipt of vaccine of SARS-CoV, MERS-CoV, SARS-CoV-2.
23. Receipt of adenovirus vector based vaccine.
24. Chronic use of immunosuppressant or immune modifying drug within 6 months prior to vaccination. (use of inhaled, topical, nasal, and ophthalmic corticosteroids are allowed)
25. Having relied on antipsychotic drugs and narcotic analgesics within 6 months before vaccination or difficult to comply with the clinical trial procedure at the judgment of the investigator.
26. Administered to other investigational product or medical device within 6 months before vaccination.
27. Other vaccination history within 30 days prior to vaccination or being scheduled within 30 days after vaccination.
28. Receipt of immunoglobulin or any blood product within 3 month prior to vaccination.
29. Pregnant(including positive hCG test at screening visit) or breastfeeding female.
30. Current smoker or vaper. (use of cigarette or e-cigarette at least once in last 30 days, Part A only)
31. Those who are directly related to the investigator.
32. Other condition deemed ineligible for the study at the discretion of investigator.

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2020-12-29 (Actual); Primary Completion 2021-07-09 (Actual); Study Completion 2023-03-27 (Actual)

PRIMARY OUTCOMES:
Incidence of solicited adverse events(AEs) | Through 7 days post-vaccination
Incidence of unsolicited AEs | Through 28, 56 days post-vaccination

SECONDARY OUTCOMES:
Incidence of serious adverse events(SAEs) | Through 12 months post-vaccination
Incidence of adverse events of special interest(AESIs) | Through 12 months post-vaccination
Seroconversion rate(SCR) of neutralization antibody using wild type SARS-CoV-2 | 4, 8 weeks post-vaccination
Geometric mean titer(GMT) of neutralization antibody using wild type SARS-CoV-2 | 4, 8 weeks post-vaccination
GMT of S protein specific antibody | 2, 4, 8, 26, 52 weeks post-vaccination
Index of T cell response | 2, 4, 26, 52 weeks post-vaccination

OTHER OUTCOMES:
SCR of neutralization antibody using pseudovirus | 2, 4, 8, 26, 52 weeks post-vaccination
GMT of neutralization antibody using pseudovirus | 2, 4, 8, 26, 52 weeks post-vaccination
GMT of S protein receptor binding domain(RBD) specific antibody | 2, 4, 8, 26, 52 weeks post-vaccination

CONTACTS AND LOCATIONS:
Locations (5):
- South Korea (5):
  - Korea University Ansan Hospital, Ansan, Province
  - The Catholic University of Korea, ST. Vincent's Hospital, Suwon, Province
  - Hallym University Kangnam Sacred Heart Hospital, Seoul, State
  - The Catholic University of Korea, Seoul ST. Mary's Hospital, Seoul, State
  - Korea University Guro Hospital, Seoul